CLINICAL TRIAL: NCT04816721
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, 2-PART STUDY TO EVALUATE EDP-938 REGIMENS IN SUBJECTS AGED 28 DAYS TO 36 MONTHS INFECTED WITH RESPIRATORY SYNCYTIAL VIRUS (RSV)
Brief Title: A Study to Evaluate EDP 938 Regimens in Children With RSV
Acronym: RSVPEDs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP 938-201
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Respiratory Syncytial Virus, RSV, Pediatric study
MeSH Terms: interventions — EDP-938

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-938 (Experimental): EDP-938, oral suspension, once daily for 5 days
  Interventions: Drug: EDP-938
- Placebo (Placebo Comparator): Matching placebo, orally, once daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 — Oral suspension
  Arms: EDP-938
Drug: Placebo — Placebo oral suspension to match EDP-938
  Arms: Placebo

SUMMARY:
A 2-part study to evaluate the safety, pharmacokinetics and efficacy of EDP-938 in children with RSV infection.

DETAILED DESCRIPTION:
This is a randomized, double-blind, dose ranging, placebo-controlled study in respiratory syncytial virus (RSV) among hospitalized and non-hospitalized children aged from 28 days to 36 months, assessing the safety, tolerability, pharmacokinetics, clinical outcome and antiviral activity of a 5 day treatment with EDP-938.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is either ≥6 months to ≤36 months (for Age Group 1) or ≥28 days to <6 months (for Age Group 2), defined at the time of randomization. Subjects in Age Group 2 must have been born ≥29 weeks of gestation to be eligible.
* Subjects diagnosed with RSV infection
* Subjects with signs of an acute respiratory illness with onset ≤7 days for Part 1 and ≤5 days for Part 2 before the time of signing the ICF
* In the Investigator's opinion, the subject's caregiver understands and is able to comply with protocol requirements, instructions, and protocol-stated restrictions, and the subject is likely to complete the study as planned

Exclusion Criteria:

* Use of or anticipated need for invasive mechanical ventilation, cardiopulmonary bypass, hemodialysis, or extracorporeal membrane oxygenation; or subjects who are not expected to survive the current illness
* Underlying immune deficiency, (e.g., from confirmed human immunodeficiency virus infection or use of an immunosuppressive medication except immunoglobulin A deficiency)
* Receipt of (within 12 months before Screening) or on a waiting list for a bone marrow, stem cell, or solid organ transplant, or who received radiation or chemotherapy (within 12 months before screening)
* Receiving chronic oxygen therapy at home before admission
* Subjects whose mother received an investigational RSV vaccination while pregnant with the subject if they were born at term (≥37 weeks of gestation) and are less than 12 months of age
* In Part 2, subjects dosed with an investigational or approved medication that is intended to prevent or treat RSV infection within the following times before the first dose of study drug: ribavirin 35 days; palivizumab 100 days; nirsevimab 350 days; other RSV-specific monoclonal antibody 5 half-lives of the specific antibody; RSV vaccines 12 months.

Ages: 28 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (78):
- United States (16):
  - Memorial Care Miller Children's and Women's Hospital, Long Beach, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California Davis, Sacramento, California
  - Nemours Children's Hospital, Orlando, Florida
  - South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Rexburg Pediatrics, Rexburg, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Norton Children's Research Institute, Louisville, Kentucky
  - MedPharmics - Lafayette, Lafayette, Louisiana
  - LSU Health, Shreveport, Louisiana
  - Willis-Knighton Health System, Shreveport, Louisiana
  - Boston Children's Hospital - Division of Adolescent/Youth Adult Medicine, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Children's Health Specialty Center Dallas Campus, Dallas, Texas
- Argentina (5):
  - Clinica del Niño y la Familia, Mar del Plata, Buenos Aires
  - Hospital Interzonal Dr Jose Penna, Bahía Blanca
  - Clínica Privada del Sol, Buenos Aires
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Clinica Central S.A, Villa Regina
- Australia (3):
  - Sydney Children's Hospital - Randwick, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Gold Coast University Hospital, Southport
- Brazil (5):
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia Hospital - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal do Paraná - Hospital de Clínicas, Curitiba
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
- Germany (3):
  - Universitätsklinikum Gießen und Marburg - Gießen, Marburg, Bundesland
  - Universitätsklinikum Erlangen, Erlangen
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah University Hospital Mount Scopu, Jerusalem
  - Schneider Children's Medical Center Of Israel, Petah Tikva
- Mexico (7):
  - Panamerican Clinical Research Mexico - Guadalajara, Guadalajara, Prados
  - Instituto Nacional de Pediatría, Mexico City
  - Hospital Infantil De Mexico Federico Gomez, Mexico City
  - Karla Adriana Espinosa Bautista, Mexico City
  - IESCI Clinical Research, Monterrey
  - PanAmerican Clinical Research, Querétaro
  - SMIQ S de R.L de C.V, Querétaro
- Wellington Regional Hospital, Newtown, Wellington Region, New Zealand
- Poland (2):
  - IN-VIVO Bydgoszcz, Bydgoszcz
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz
- Romania (3):
  - Spital Clinic de Urgenta Pentru Copii Brasov, Brasov, Brașov County
  - Spitalul Clinic Judetean De Urgenta Târgu Mureș, Târgu Mureş, Târgu Mureș
  - Institutul National pentru Sanatatea Mamei si Copilului "Alessandrescu-Rusescu", Bucharest
- South Africa (3):
  - Life Westville Hospital, Westville, Durban
  - Rahima Moosa Mother and Child Hospital, Johannesburg
  - Wits Clinical Research, Soweto
- South Korea (3):
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kyung Hee University Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
- Spain (13):
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
  - Unidad de Ensayos Clínicos Pediátricos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Joan XXIII de Tarragona, Tarragona
- Taiwan (6):
  - National Taiwan University Hospital, Taipei City, Taipei
  - Linkou Chang Gung Memorial Hospital, Chang Gung Medical Foundation, Taoyuan, Taoyuan
  - Hsinchu Mackay Memorial Hospital, Hsinchu
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Mackay Memorial Hospital, Taipei
- United Kingdom (3):
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - St. George's University Hospitals NHS Foundation Trust, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 99 participants were enrolled at 78 sites across 15 countries between April 2022 and August 2024.
Pre-assignment Details: Participants were randomized 2:1 (Part 1) or 4:1 (Part 2) to EDP-938:placebo.
Groups:
- Part 1, Group 1: EDP-938: Participants aged ≥ 6 months to < 12 months received oral 5 mg/kg doses of EDP-938 once daily (QD) from Day 1 to Day 5 of the study. Participants aged ≥ 12 months to ≤ 36 months received oral 5 mg/kg or 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1, Group 2: EDP-938; Part 2, Group 2: EDP-938: Participants aged ≥ 28 days to < 6 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1, Group 1: Placebo: Participants aged ≥ 6 months to ≤ 36 months received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1, Group 2: Placebo; Part 2, Group 2: Placebo: Participants aged between ≥ 28 days and < 6 months received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2, Group 1: EDP-938: Participants aged ≥ 6 months to < 12 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study. Participants aged ≥ 12 months to ≤ 36 months received oral 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2, Group 1: Placebo: Participants aged between ≥ 6 months and ≤ 36 months received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
Period: Overall Study
Arm/Group | Part 1, Group 1: EDP-938 | Part 1, Group 2: EDP-938 | Part 1, Group 1: Placebo | Part 1, Group 2: Placebo | Part 2, Group 1: EDP-938 | Part 2, Group 2: EDP-938 | Part 2, Group 1: Placebo | Part 2, Group 2: Placebo
Started | 22 | 14 | 11 | 6 | 20 | 16 | 6 | 4
Treated With 5 mg/kg EDP-938 | 14 | 13 | 0 | 0 | 8 | 15 | 0 | 0
Treated With 7.5 mg/kg EDP-938 (1 participant was randomized to placebo, but received 7.5 mg/kg EDP-938 in error.) | 9 | 0 | 0 | 0 | 11 | 0 | 0 | 0
Treated With Placebo | 0 | 0 | 11 | 6 | 0 | 0 | 6 | 4
Completed | 22 | 12 | 11 | 4 | 19 | 15 | 6 | 4
Not Completed | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Included all participants who received any dose (including partial doses) of any study drug. Participants have been reported according to the actual treatment received. One participant was randomized to 7.5 mg/kg EDP-938, but received 5 mg/kg in error and one participant was randomized to placebo, but received 7.5 mg/kg EDP-938 in error.
Groups:
- Part 1, Group 1: EDP-938: Participants aged ≥ 6 months to < 12 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study. Participants aged ≥ 12 months to ≤ 36 months received oral 5 mg/kg or 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1, Group 1: Placebo; Part 2, Group 1: Placebo: Participants aged between ≥ 6 months and ≤ 36 months received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1, Group 1: EDP-938 | Part 1, Group 2: EDP-938 | Part 1, Group 1: Placebo | Part 1, Group 2: Placebo | Part 2, Group 1: EDP-938 | Part 2, Group 2: EDP-938 | Part 2, Group 1: Placebo | Part 2, Group 2: Placebo | Total
Number analyzed (Participants) | 23 | 13 | 10 | 6 | 19 | 15 | 6 | 4 | 96
Age, Customized [Count of Participants; unit: Participants]
  ≥ 28 days to < 3 months | 0 | 9 | 0 | 4 | 0 | 7 | 0 | 2 | 22
  ≥ 3 months to < 6 months | 0 | 4 | 0 | 2 | 0 | 8 | 0 | 2 | 16
  ≥ 6 months to < 12 months | 7 | 0 | 4 | 0 | 8 | 0 | 3 | 0 | 22
  ≥ 12 months to ≤ 36 months | 16 | 0 | 6 | 0 | 11 | 0 | 3 | 0 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 3 | 5 | 11 | 7 | 5 | 1 | 49
  Male | 11 | 8 | 7 | 1 | 8 | 8 | 1 | 3 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 3 | 3 | 2 | 6 | 6 | 3 | 3 | 38
  Not Hispanic or Latino | 11 | 10 | 7 | 4 | 12 | 9 | 3 | 1 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 9
  Black or African American | 3 | 0 | 5 | 2 | 3 | 2 | 0 | 0 | 15
  White | 18 | 11 | 3 | 2 | 12 | 10 | 4 | 2 | 62
  Other | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 6
  Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hospitalization Status on Day 1 [Count of Participants; unit: Participants]
  Yes | 16 | 12 | 8 | 5 | 17 | 12 | 4 | 3 | 77
  No | 7 | 1 | 2 | 1 | 2 | 3 | 2 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Concentrations of EDP-938 in Plasma
Description: Plasma concentrations of EDP-938 were assessed at the designated time points.
Time Frame: 3 hours post-dose on Day 1 and pre-dose on Day 2 (hospitalized participants only), Day 3, and Day 5
Population: Pharmacokinetic (PK) Population: Included all participants in Part 1 who received one full dose of study drug and had samples with quantifiable plasma levels to allow for estimation of PK parameters. Per protocol, data were analyzed per age group and dose received.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1: EDP-938 5mg/kg (≥ 28 Days to < 3 Months): Participants aged between ≥ 28 days and < 3 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1: EDP-938 5mg/kg (≥ 3 Months to < 6 Months): Participants aged between ≥ 3 months and < 6 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1: EDP-938 5mg/kg (≥ 6 Months to < 12 Months): Participants aged between ≥ 6 months and < 12 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1: EDP-938 5mg/kg (≥ 12 Months to ≤ 36 Months): Participants aged between ≥ 12 months to ≤ 36 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1: EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months): Participants aged between ≥ 12 months to ≤ 36 months received oral 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Part 1: EDP-938 5mg/kg (≥ 28 Days to < 3 Months) | Part 1: EDP-938 5mg/kg (≥ 3 Months to < 6 Months) | Part 1: EDP-938 5mg/kg (≥ 6 Months to < 12 Months) | Part 1: EDP-938 5mg/kg (≥ 12 Months to ≤ 36 Months) | Part 1: EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months)
Number analyzed (Participants) | 9 | 4 | 7 | 7 | 9
ng/mL
  Day 1: number analyzed (Participants) | 9 | 4 | 7 | 6 | 8
  Day 1 | 1132.222 (397.4289) | 1989.500 (1331.5646) | 1819.286 (809.9508) | 1420.000 (604.8140) | 1428.250 (817.4801)
  Day 2: number analyzed (Participants) | 7 | 4 | 4 | 4 | 7
  Day 2 | 368.400 (149.8741) | 399.250 (423.9515) | 502.350 (379.6487) | 249.675 (294.5416) | 238.900 (239.0287)
  Day 3: number analyzed (Participants) | 2 | 0 | 3 | 3 | 2
  Day 3 | 448.000 (229.1026) |  | 346.000 (54.7449) | 97.533 (64.9043) | 116.250 (43.4871)
  Day 5: number analyzed (Participants) | 7 | 4 | 7 | 7 | 9
  Day 5 | 528.563 (284.6010) | 201.750 (98.6623) | 431.429 (637.5664) | 252.043 (329.2155) | 180.622 (158.3268)

2. Primary Outcome: Part 1: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were defined as any event, side effect, or untoward medical occurrence in a participant enrolled in a clinical study whether or not it was considered to have a causal relationship to the study drug and first occurred or worsened during the post-baseline phase compared to baseline. Clinically significant changes from baseline in vital signs and clinical laboratory results were reported as TEAEs.
Time Frame: Day 1 to Day 28
Population: Safety Population: Included all participants in Part 1 who received any dose (including partial doses) of any study drug. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: EDP-938: Participants who received oral doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 1: Placebo: Participants who received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Part 1: EDP-938 | Part 1: Placebo
Number analyzed (Participants) | 36 | 16
Participants | 14 | 9

3. Primary Outcome: Part 2: Model-Adjusted Daily Change From Baseline in Respiratory Syncytial Virus (RSV) Shedding in Nasal Swab Samples
Description: Daily change from baseline in RSV shedding was defined as the daily change from baseline in RSV ribonucleic acid (RNA) viral load and was measured using reverse transcription-quantitative polymerase chain reaction (RT-qPCR) from nasal swabs. The model included treatment group (EDP-938, placebo) and Day (3, 5, 9, and 14) as fixed effect, associated baseline, and treatment group by Day interaction term as factors. An unstructured covariance matrix was imposed. The Satterthwaite approximation is used to estimate the denominator degrees of freedom.
Time Frame: Baseline and pre-dose on Days 3, 5, 9, and 14
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Groups:
- Part 2: EDP-938: Participants who received oral doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2: Placebo: Participants who received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 34 | 10
log10 copies/mL
  Day 3 | -1.33 (0.297) | -0.37 (0.533)
  Day 5 | -3.04 (0.354) | -1.62 (0.627)
  Day 9 | -3.65 (0.381) | -3.22 (0.680)
  Day 14 | -4.87 (0.388) | -5.71 (0.677)
Statistical Analysis 1: Comparison: Part 2: EDP-938 vs Part 2: Placebo; Day 3: EDP-938 Versus Placebo; Test type: Superiority — The model included treatment group (EDP-938, placebo) and Day (3, 5, 9, and 14) as fixed effect, associated baseline, and treatment group by day interaction term as factors. An unstructured covariance matrix was imposed. The Satterthwaite approximation was used to estimate the denominator degrees of freedom; p = 0.1249, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.96, 95% CI 2-sided [-2.21 to 0.28]
Statistical Analysis 2: Comparison: Part 2: EDP-938 vs Part 2: Placebo; Day 5: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0580, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -1.41, 95% CI 2-sided [-2.88 to 0.05]
Statistical Analysis 3: Comparison: Part 2: EDP-938 vs Part 2: Placebo; Day 9: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.5877, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.43, 95% CI 2-sided [-2.02 to 1.16]
Statistical Analysis 4: Comparison: Part 2: EDP-938 vs Part 2: Placebo; Day 14: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.2932, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = 0.84, 95% CI 2-sided [-0.76 to 2.43]

4. Primary Outcome: Pooled Population: Model-Adjusted Daily Change From Baseline in RSV Shedding in Nasal Swab Samples
Description: Daily change from baseline in RSV shedding was defined as the daily change from baseline in RSV RNA viral load and was measured using RT-qPCR from nasal swabs. The model included treatment group (EDP-938, placebo) and Day (3, 5, 9, and 14) as fixed effect, associated baseline, and treatment group by Day interaction term as factors. An unstructured covariance matrix was imposed.The Satterthwaite approximation is used to estimate the denominator degrees of freedom.
Time Frame: Baseline and pre-dose on Days 3, 5, 9, and 14
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Groups:
- Combined EDP-938: Participants in Part 1 and Part 2 who received oral doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Combined Placebo: Participants in Part 1 and Part 2 who received oral doses of placebo matching EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 69 | 27
log10 copies/mL
  Day 3 | -1.53 (0.192) | -1.36 (0.331)
  Day 5 | -2.95 (0.230) | -2.62 (0.392)
  Day 9 | -4.57 (0.275) | -3.87 (0.475)
  Day 14 | -5.01 (0.278) | -5.35 (0.462)
Statistical Analysis 1: Comparison: Combined EDP-938 vs Combined Placebo; Day 3: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.6574, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.93 to 0.59]
Statistical Analysis 2: Comparison: Combined EDP-938 vs Combined Placebo; Day 5: EDP-938 Versus Placebo; Test type: Superiority; p = 0.4728, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-1.23 to 0.58]
Statistical Analysis 3: Comparison: Combined EDP-938 vs Combined Placebo; Day 9: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.2058, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-1.79 to 0.39]
Statistical Analysis 4: Comparison: Combined EDP-938 vs Combined Placebo; Day 14: EDP-938 Versus Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.5391, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = 0.33, 95% CI 2-sided [-0.74 to 1.41]

5. Secondary Outcome: Part 1 and Part 2: Area Under the Curve (AUC) for RSV RNA Viral Load
Description: The RSV RNA viral load was measured using RT-qPCR from nasal swabs. The AUC was calculated using the trapezoid rule. The AUC was calculated based on all available assessments collected on Days 1, 3, 5, 9 and 14 and the actual date/time of each assessment was used for the calculation.
Time Frame: Pre-dose on Day 1 through pre-dose on Days 3, 5, 9 and 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 copies/mL*Days
Arm/Group | Part 1: EDP-938 | Part 1: Placebo | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 34 | 12 | 29 | 9
log10 copies/mL*Days
  Day 1 through Day 3: number analyzed (Participants) | 34 | 12 | 25 | 9
  Day 1 through Day 3 | 17.80 (4.522) | 17.26 (4.691) | 17.15 (4.663) | 16.91 (3.266)
  Day 1 through Day 5 | 25.54 (8.301) | 24.55 (8.457) | 24.76 (7.914) | 26.22 (7.069)
  Day 1 through Day 9 | 36.03 (16.229) | 35.20 (17.156) | 37.00 (13.652) | 40.39 (13.371)
  Day 1 through Day 14 | 42.85 (24.990) | 44.16 (25.056) | 45.49 (21.109) | 42.17 (19.864)

6. Secondary Outcome: Pooled Population: AUC of Change From Baseline in RSV RNA Viral Load
Description: The RSV RNA viral load was measured using RT-qPCR from nasal swabs. The AUC was calculated using the trapezoid rule. The AUC was calculated based on all available assessments collected on Days 1, 3, 5, 9 and 14 and the actual date/time of each assessment was used for the calculation. The model included treatment group (EDP-938, placebo) and Day (3, 5, 9, and 14) as fixed effect, associated baseline, and treatment group by day interaction term as factors. An unstructured covariance matrix was imposed. The Satterthwaite approximation was used to estimate the denominator degrees of freedom.
Time Frame: Baseline (Pre-dose on Day 1) through pre-dose on Days 3, 5, 9 and 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL*Days
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 69 | 27
log10 copies/mL*Days
  Day 1 through Day 3 | -1.53 (0.192) | -1.36 (0.331)
  Day 1 through Day 5 | -6.00 (0.540) | -5.33 (0.930)
  Day 1 through Day 9 | -21.04 (1.319) | -18.32 (2.272)
  Day 1 through Day 14 | -45.00 (2.105) | -41.36 (3.619)
Statistical Analysis 1: Comparison: Combined EDP-938 vs Combined Placebo; Day 1 through Day 3: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.6574, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.93 to 0.59]
Statistical Analysis 2: Comparison: Combined EDP-938 vs Combined Placebo; Day 1 through Day 5: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.5359, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -0.67, 95% CI 2-sided [-2.81 to 1.47]
Statistical Analysis 3: Comparison: Combined EDP-938 vs Combined Placebo; Day 1 through Day 9: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.3029, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -2.73, 95% CI 2-sided [-7.95 to 2.50]
Statistical Analysis 4: Comparison: Combined EDP-938 vs Combined Placebo; Day 1 through Day 14: EDP-938 Versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.3871, Mixed-effect Model of Repeated Measures; Least Squares Mean Difference = -3.64, 95% CI 2-sided [-11.98 to 4.69]

7. Secondary Outcome: Part 1: Daily Change From Baseline in RSV Shedding in Nasal Swab Samples
Description: Daily change from baseline in RSV shedding in nasal swab samples was defined as the absolute daily change from baseline in RSV RNA viral load and measured using RT-qPCR from nasal swabs.
Time Frame: Baseline to pre-dose on Days 3, 5, 9, and Day 14
Population: Efficacy Population: Included all participants in Part 1 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part 1: EDP-938 | Part 1: Placebo
Number analyzed (Participants) | 34 | 12
log10 copies/mL
  Day 3 | -1.68 (1.239) | -2.17 (1.948)
  Day 5: number analyzed (Participants) | 33 | 12
  Day 5 | -2.91 (1.634) | -3.44 (1.585)
  Day 9: number analyzed (Participants) | 32 | 11
  Day 9 | -5.34 (2.338) | -4.41 (1.897)
  Day 14: number analyzed (Participants) | 31 | 12
  Day 14 | -5.11 (2.378) | -5.15 (2.118)

8. Secondary Outcome: Part 1 and Part 2: Percentage of Participants With RSV RNA Viral Load Below the Limit of Detection (LOD)
Description: The RSV RNA viral load was measured using RT-qPCR from nasal swabs.
Time Frame: Pre-dose on Days 3, 5, 9 and 14
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Included only participants with detectable viral load at baseline and non-missing viral load assessment at the respective visit and was used as a denominator in the percentage population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: EDP-938 | Part 1: Placebo | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 34 | 12 | 28 | 9
percentage of participants
  Day 3 | 0 [0.00 to 10.28] | 8.3 [0.21 to 38.48] | 3.6 [0.09 to 18.35] | 0 [0.00 to 33.63]
  Day 5: number analyzed (Participants) | 33 | 12 | 27 | 9
  Day 5 | 12.1 [3.40 to 28.20] | 16.7 [2.09 to 48.41] | 22.2 [8.62 to 42.26] | 0 [0.00 to 33.63]
  Day 9: number analyzed (Participants) | 32 | 11 | 25 | 8
  Day 9 | 62.5 [43.69 to 78.90] | 36.4 [10.93 to 69.21] | 28.0 [12.07 to 49.39] | 25.0 [3.19 to 65.09]
  Day 14: number analyzed (Participants) | 31 | 12 | 27 | 9
  Day 14 | 61.3 [42.19 to 78.15] | 58.3 [27.67 to 84.83] | 63.0 [42.37 to 80.60] | 88.9 [51.75 to 99.72]

9. Secondary Outcome: Pooled Population: Percentage of Participants With RSV RNA Viral Load Below the LOD
Description: The RSV RNA viral load was measured using RT-qPCR from nasal swabs.
Time Frame: Pre-dose on Days 3, 5, 9 and 14
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 62 | 21
percentage of participants
  Day 3 | 1.6 [0.04 to 8.66] | 4.8 [0.12 to 23.82]
  Day 5: number analyzed (Participants) | 60 | 21
  Day 5 | 16.7 [8.29 to 28.52] | 9.5 [1.17 to 30.38]
  Day 9: number analyzed (Participants) | 57 | 19
  Day 9 | 47.4 [33.98 to 61.03] | 31.6 [12.58 to 56.55]
  Day 14: number analyzed (Participants) | 58 | 21
  Day 14 | 62.1 [48.37 to 74.49] | 71.4 [47.82 to 88.72]

10. Secondary Outcome: Part 1 and Part 2: Time to RSV RNA Viral Load Being Undetectable
Description: Time to RSV RNA viral load being undetectable was calculated as: first date of RSV RNA viral load target not detected (TND) after which no further samples had detectable RSV RNA viral load - date of first dose.
Time Frame: Day 1 to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 1: EDP-938 | Part 1: Placebo | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 34 | 14 | 29 | 9
days | 10.59 (3.661) | 12.33 (3.018) | 12.46 (3.235) | 12.19 (3.040)

11. Secondary Outcome: Pooled Population: Time to RSV RNA Viral Load Being Undetectable
Description: Time to RSV RNA viral load being undetectable was calculated as: first date of RSV RNA viral load TND after which no further samples had detectable RSV RNA viral load - date of first dose.
Time Frame: Day 1 to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 63 | 23
days | 11.45 (3.570) | 12.27 (2.958)

12. Secondary Outcome: Part 2: Number of Participants Who Experienced a TEAE
Description: as for outcome 2
Time Frame: Day 1 to Day 28
Population: Safety Population: Included all participants in Part 2 who received any dose (including partial doses) of any study drug. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 34 | 10
Participants | 14 | 4

13. Secondary Outcome: Pooled Population: Number of Participants Who Experienced a TEAE
Description: as for outcome 2
Time Frame: Day 1 to Day 28
Population: Safety Population: Included all participants who received any dose (including partial doses) of any study drug. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 70 | 26
Participants | 28 | 13

14. Secondary Outcome: Part 2: Concentrations of EDP-938 in Plasma
Description: Plasma concentrations of EDP-938 were assessed at the designated time points.
Time Frame: 3 hours post-dose on Day 1 and pre-dose on Day 2 (hospitalized participants only), Day 3, and Day 5
Population: PK Population: Included all participants in Part 2 who received one full dose of study drug and had samples with quantifiable plasma levels to allow for estimation of PK parameters. Per protocol, data were analyzed per age group and dose received.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 2: EDP-938 5mg/kg (≥ 28 Days to < 3 Months): Participants aged between ≥ 28 days and < 3 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2: EDP-938 5mg/kg (≥ 3 Months to < 6 Months): Participants aged between ≥ 3 months and < 6 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2: EDP-938 5mg/kg (≥ 6 Months to < 12 Months): Participants aged between ≥ 6 months and < 12 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Part 2: EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months): Participants aged between ≥ 12 months to ≤ 36 months received oral 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Part 2: EDP-938 5mg/kg (≥ 28 Days to < 3 Months) | Part 2: EDP-938 5mg/kg (≥ 3 Months to < 6 Months) | Part 2: EDP-938 5mg/kg (≥ 6 Months to < 12 Months) | Part 2: EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months)
Number analyzed (Participants) | 7 | 8 | 7 | 9
ng/mL
  Day 1 | 1116.286 (217.9983) | 1169.903 (802.0744) | 1551.429 (363.8419) | 1368.111 (469.7815)
  Day 2: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 2 | 585.400 (119.6089) | 273.500 (150.4616) | 140.783 (73.3099) | 200.700 (134.3896)
  Day 3: number analyzed (Participants) | 1 | 2 | 1 | 3
  Day 3 | 194.000 (NA) — Standard deviation was not estimable as only 1 participant had available data. | 926.000 (57.9828) | 112.000 (NA) — Standard deviation was not estimable as only 1 participant had available data. | 115.967 (84.9347)
  Day 5: number analyzed (Participants) | 6 | 7 | 7 | 8
  Day 5 | 516.333 (247.6697) | 519.714 (436.8130) | 69.110 (40.4604) | 153.450 (102.4372)

15. Secondary Outcome: Pooled Population: Concentrations of EDP-938 in Plasma
Description: Plasma concentrations of EDP-938 were assessed at the designated time points.
Time Frame: 3 hours post-dose on Day 1 and pre-dose on Day 2 (hospitalized participants only), Day 3, and Day 5
Population: PK Population: Included all participants who received one full dose of study drug and had samples with quantifiable plasma levels to allow for estimation of PK parameters. Per protocol, data were analyzed per age group and dose received.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Combined EDP-938 5mg/kg (≥ 28 Days to < 3 Months): Participants aged between ≥ 28 days and < 3 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Combined EDP-938 5mg/kg (≥ 3 Months to < 6 Months): Participants aged between ≥ 3 months and < 6 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Combined EDP-938 5mg/kg (≥ 6 Months to < 12 Months): Participants aged between ≥ 6 months and < 12 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Combined EDP-938 5mg/kg (≥ 12 Months to ≤ 36 Months): Participants aged between ≥ 12 months to ≤ 36 months received oral 5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
- Combined EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months): Participants aged between ≥ 12 months to ≤ 36 months received oral 7.5 mg/kg doses of EDP-938 QD from Day 1 to Day 5 of the study.
Arm/Group | Combined EDP-938 5mg/kg (≥ 28 Days to < 3 Months) | Combined EDP-938 5mg/kg (≥ 3 Months to < 6 Months) | Combined EDP-938 5mg/kg (≥ 6 Months to < 12 Months) | Combined EDP-938 5mg/kg (≥ 12 Months to ≤ 36 Months) | Combined EDP-938 7.5 mg/kg (≥ 12 Months to ≤ 36 Months)
Number analyzed (Participants) | 16 | 12 | 14 | 7 | 18
ng/mL
  Day 1: number analyzed (Participants) | 16 | 12 | 14 | 6 | 17
  Day 1 | 1125.250 (321.4278) | 1443.102 (1027.5197) | 1685.357 (619.0267) | 1420.000 (604.8140) | 1396.412 (635.3537)
  Day 2: number analyzed (Participants) | 12 | 10 | 10 | 4 | 13
  Day 2 | 458.817 (173.0322) | 323.800 (276.9576) | 285.410 (293.0727) | 249.675 (294.5416) | 221.269 (191.0117)
  Day 3: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5
  Day 3 | 363.333 (218.5162) | 926.000 (57.9828) | 287.500 (125.2478) | 97.533 (64.9043) | 116.080 (63.8730)
  Day 5: number analyzed (Participants) | 13 | 11 | 14 | 7 | 17
  Day 5 | 522.918 (257.0945) | 404.091 (378.3365) | 250.269 (472.9799) | 252.043 (329.2155) | 167.835 (131.6054)

16. Secondary Outcome: Part 2: Time to First Hospital Discharge for Hospitalized Participants
Description: Time to first discharge for participants who were hospitalized at randomization was calculated as: date/time of first discharge - date/time of first dose with conversion to days. For participants with continuous hospitalization, the last date of discharge from the continuous hospitalization was used.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Only participants who were hospitalized at randomization were included. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 29 | 7
days | 3.93 (1.870) | 4.00 (3.367)

17. Secondary Outcome: Pooled Population: Time to First Hospital Discharge for Hospitalized Participants
Description: as for outcome 16
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Only participants who were hospitalized at randomization were included. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 56 | 21
days | 3.71 (2.006) | 3.57 (2.959)

18. Secondary Outcome: Part 2: Time to Use of Oxygen for Hospitalized Participants Who Were Not Receiving Oxygen at the Time They Received the First Dose of Study Drug
Description: For participants were were hospitalized at randomization, time to use of oxygen for hospitalization participants who were not receiving oxygen at the time they received the first dose of study drug was calculated as: first date/time of receiving oxygen - date/time of first dose of study drug with conversion to days.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. As there were no participants in Part 2 in both arms who were hospitalized at randomization who were not receiving oxygen at the time they received the first dose of study drug, no data were collected for this outcome measure.
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Pooled Population: Time to Use of Oxygen for Hospitalized Participants Who Were Not Receiving Oxygen at the Time They Received the First Dose of Study Drug
Description: as for outcome 18
Time Frame: Day 1 to Day 28
Population: Efficacy Population. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only hospitalized participants who were not receiving oxygen at the time they received the first dose of study drug were included. In the Placebo arm, there were no hospitalized participants who were not receiving oxygen at the time they received the first dose of study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 1 | 0
days | 0.51 (NA) — Standard deviation was not estimable as only 1 participant had available data. |

20. Secondary Outcome: Part 2: Percentage of Hospitalized Participants Who Required Oxygen Supplementation or Had an Increased Oxygen Requirement After the First Dose of Study Drug
Description: The numerator in the percentage calculation was defined by the number of participants who developed a new requirement for oxygen supplementation or new increase in oxygen requirements after the first dose of study drug, based on the response of "yes" to the "Is this an increase of oxygen supplementation compared to previous use?" question on the Oxygen Supplementation case report form (CRF). The 95% confidence interval was reported using the Clopper Pearson confidence interval methods.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were hospitalized at randomization and/or during the study were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 29 | 7
percentage of participants | 24.1 [10.30 to 43.54] | 28.6 [3.67 to 70.96]

21. Secondary Outcome: Pooled Population: Percentage of Hospitalized Participants Who Required Oxygen Supplementation or Had an Increased Oxygen Requirement After the First Dose of Study Drug
Description: The numerator in the percentage calculation was defined by the number of participants who developed a new requirement for oxygen supplementation or new increase in oxygen requirements after the first dose of study drug, based on the response of "yes" to the "Is this an increase of oxygen supplementation compared to previous use?" question on the Oxygen Supplementation CRF. The 95% confidence interval was reported using the Clopper Pearson confidence interval methods.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were hospitalized at randomization and/or during the study were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 56 | 21
percentage of participants | 25.0 [14.39 to 38.37] | 19.0 [5.45 to 41.91]

22. Secondary Outcome: Part 2: Time to Mechanical Ventilation for Hospitalized Participants
Description: Time to mechanical ventilation for participants who were hospitalized at randomization was calculated as: first date/time of mechanical ventilation - date/time of first dose of study drug with conversion to days. Participants who were on mechanical ventilation before their first dose of study drug were excluded from the analysis.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. As only participants who were hospitalized at baseline and experienced mechanical ventilation were included, no data were collected for this outcome measure.
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Pooled Population: Time to Mechanical Ventilation for Hospitalized Participants
Description: as for outcome 22
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. As only participants who were hospitalized at baseline and experienced mechanical ventilation after their first dose of study drug were included, no data were collected for this outcome measure.
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part 2: Percentage of Hospitalized Participants Who Required Mechanical Ventilation
Description: The numerator in the percentage calculation was defined by the number of participants who developed a new requirement for mechanical ventilation after the first dose of study drug. Participants on mechanical ventilation prior to the first dose of study drug were excluded from analysis. The 95% confidence interval was reported using the Clopper Pearson confidence interval methods.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only hospitalized participants who were not on mechanical ventilation prior to the first dose of study drug were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 29 | 7
percentage of participants | 0 [0.00 to 11.94] | 0 [0.00 to 40.96]

25. Secondary Outcome: Pooled Population: Percentage of Hospitalized Participants Who Required Mechanical Ventilation
Description: as for outcome 24
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only hospitalized participants who were not on mechanical ventilation prior to the first dose of study drug were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 56 | 21
percentage of participants | 0 [0.00 to 6.38] | 0 [0.00 to 16.11]

26. Secondary Outcome: Part 2: Percentage of Hospitalized Participants Who Died During the Study
Description: The percentage of hospitalized participants who died during the study included deaths from any cause. The 95% confidence interval was reported using the Clopper Pearson confidence interval methods.
Time Frame: Day 1 to Day 28
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 29 | 7
percentage of participants | 0 [0.00 to 11.94] | 0 [0.00 to 40.96]

27. Secondary Outcome: Pooled Population: Percentage of Hospitalized Participants Who Died During the Study
Description: as for outcome 26
Time Frame: Day 1 to Day 28
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 56 | 21
percentage of participants | 0 [0.00 to 6.38] | 0 [0.00 to 16.11]

28. Secondary Outcome: Part 2: Time to Hospitalization for Initial Outpatients Who Were Subsequently Hospitalized
Description: Time to hospitalization for initial outpatients who are not hospitalized at randomization but subsequently hospitalized was calculated as: first date/time of hospitalization - date/time of first dose with conversion to days.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. As only participants who were not hospitalized at randomization but subsequently hospitalized were included, no data were collected for this outcome measure.
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Pooled Population: Time to Hospitalization for Initial Outpatients Who Were Subsequently Hospitalized
Description: as for outcome 28
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. As only participants who were not hospitalized at randomization but subsequently hospitalized were included, no data were collected for this outcome measure.
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part 2: Percentage of Outpatients Who Were Subsequently Hospitalized or Died
Description: Participants who were hospitalized at randomization were excluded from the analysis. The 95% confidence interval was reported using the Clopper Pearson confidence interval methods.
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were not hospitalized at randomization were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 5 | 3
percentage of participants | 0 [0.00 to 52.18] | 0 [0.00 to 70.76]

31. Secondary Outcome: Pooled Population: Percentage of Outpatients Who Were Subsequently Hospitalized or Died
Description: as for outcome 30
Time Frame: Day 1 to Day 28
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were not hospitalized at randomization were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 13 | 6
percentage of participants | 0 [0.00 to 24.71] | 0 [0.00 to 45.93]

32. Secondary Outcome: Part 2: Time to Resolution of Symptoms for Outpatients Who Were Not Hospitalized
Description: Resolution of symptoms was defined as the first of 2 consecutive timepoints where each of the seven symptoms assessed by the Parent/Caregiver Respiratory Syncytial Virus (RSV) Foundation (ReSVinet) score was 0 (not present) or 1 (mild). Time to resolution of symptoms for outpatients who were not hospitalized was calculated as: first date/time of resolution of symptoms - date/time of first dose with conversion to days. Participants who did not achieve resolution and had not been followed through the Day 14 visit or completed the Day 14 questionnaire were censored at Day 14.
  During the study, the parent(s)/caregiver(s) assessed the severity of RSV-related signs and symptoms. The ReSVinet assessed 7 symptoms, with each symptom being rated from 0 (not present) to 3 (severe), apart from fever which was scored from 0-2. The full range was 0 to 20 with higher scores representing more severe disease.
Time Frame: Day 1 to Day 14
Population: Efficacy Population: Included all participants in Part 2 who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were not hospitalized were included.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 2: EDP-938 | Part 2: Placebo
Number analyzed (Participants) | 3 | 2
days | 2.60 (1.686) | 1.49 (0.702)

33. Secondary Outcome: Pooled Population: Time to Resolution of Symptoms for Outpatients Who Were Not Hospitalized
Description: Resolution of symptoms was defined as the first of 2 consecutive timepoints where each of the seven symptoms assessed by the Parent/Caregiver ReSVinet score was 0 (not present) or 1 (mild). Time to resolution of symptoms for outpatients who were not hospitalized was calculated as: first date/time of resolution of symptoms - date/time of first dose with conversion to days. Participants who did not achieve resolution and had not been followed through the Day 14 visit or completed the Day 14 questionnaire were censored at Day 14.
  During the study, the parent(s)/caregiver(s) assessed the severity of RSV-related signs and symptoms. The ReSVinet assessed 7 symptoms, with each symptom being rated from 0 (not present) to 3 (severe), apart from fever which was scored from 0-2. The full range was 0 to 20 with higher scores representing more severe disease.
Time Frame: Day 1 to Day 14
Population: Efficacy Population: Included all participants who received one full dose of study drug and had at least one evaluable measurement while on treatment. Per the protocol, analyses were planned to be grouped by EDP-938 and placebo, rather than by dose. Only participants who were not hospitalized were included.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Combined EDP-938 | Combined Placebo
Number analyzed (Participants) | 8 | 5
days | 2.42 (1.163) | 4.20 (5.552)

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: The analysis population for serious adverse events and other (non-serious) adverse events was the safety population which included all participants who received any dose (including partial doses) of any study drug. Per Section 4.1 of the SAP, analyses were planned to be grouped by treatment, rather than by specific dose.
Arm/Group | Part 1: EDP-938 | Part 1: Placebo | Part 2: EDP-938 | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/16 | 0/34 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/36 | 2/16 | 1/34 | 0/10
Other Adverse Events (participants affected / at risk) | 7/36 | 7/16 | 9/34 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: EDP-938 (N=36) | Part 1: Placebo (N=16) | Part 2: EDP-938 (N=34) | Part 2: Placebo (N=10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: EDP-938 (N=36) | Part 1: Placebo (N=16) | Part 2: EDP-938 (N=34) | Part 2: Placebo (N=10)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04816721/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT04816721/SAP_001.pdf